CLINICAL TRIAL: NCT05675891
Title: The Effect of Supplemental Feeding System on Preterm Infants' Oral Feeding Skils: Randomized Controlled Trial
Brief Title: Oral Feeding Ability of Preterm Infants With Breastfeeding Support System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Fatma BOZDAG, Lecturer Doctor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HRU-BOZDAG-001
Record Dates: First submitted 2022-12-10; First posted 2023-01-09 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Nutrition Disorder, Infant; Nutrition
Keywords: Preterm infants; Early feeding skills; Supplemental feeding system
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemental Feeding System Group (Experimental): 3 feeding between 08-16:00 are carried out with the supplemental feeding system. The remaining 5 feedings continue with the bottle.
  Interventions: Other: Supplemental Feeding System Group
- Bottle Feeding Group (Control) (No Intervention): All feedings are made from a bottle.

INTERVENTIONS:
Other: Supplemental Feeding System Group — The body weight is measured in the morning fasting on the day when oral feeding is decided, 3 feeding between 08-16:00 are carried out with the supplemental feeding system, The amount of food prepared is recorded, Heart rate, oxygen saturation, respiratory rate and early feeding skill score are recorded before, during and after feeding, When the feeding is finished, the total amount of food taken by the baby and the feeding time are recorded, The rate of food intake (%) and the amount of food received per minute are calculated and recorded, Infants who can take 80% of the amount of food given at each meal by being fed orally for 8 meals two days in a row are considered to have switched to full oral feeding.
  Arms: Supplemental Feeding System Group

SUMMARY:
This research 34.-36. is carried out as a randomized controlled experimental design in order to evaluate the effectiveness of the supplemental feeding system to improve the early feeding skills of preterm infants receiving care in the neonatal intensive care unit at the gestational week.The universe of this research will consist of preterm infants hospitalized in the neonatal intensive care of Sanlıurfa Training and Research Hospital between July 2022 and April 2023. The sample size in the study was "H00: There is no difference between preterm infants with supplemental feeding system and preterm infants fed with bottle in terms of early feeding skills." According to the hypothesis G*Power Version 3.1.9.2 (Franz Foul, Universitat Kiel, Germany) was calculated in the program. In order to determine the difference between the groups, the number of groups is 2; number of repeated measurements 3; correlation between repeated measurements 0.5; Cohen* effect size 0.25; The statistical power was determined as a sample size of 44 preterm infants, 22 of whom were fed with supplemental feeding system and 22 of whom were fed with bottle, with 95% and type 1 error of 5%. and infants assigned to groups by randomization method. Randomization in the study determined by entering the total number of cases through the program http://www.randomizer.org. Through this program, the infants forming the sample group randomly distributed to two groups and randomization made.

DETAILED DESCRIPTION:
Written and verbal consents are obtained by informing the mothers about the study, and the information about the preterm infants and their mothers is recorded. Preterm infants, whose transition to oral feeding was decided by the physician and nurse and whose families gave consent to participate in the study, were randomly assigned to 2 groups as experimental (supplemental feeding system; SFS) and control (bottle feeding group; BFG). After oral feeding is decided, the first feeding of preterm infants in both groups is tried directly on the mother's breast and the early feeding skill score is 57, with heart rate (120-160/min), sPO2(>90) and respiratory rates (40-60/min) during the time they are at the mother's breast. min) are not included in the study, whose follow-ups are between normal values. The first feeding of the infants in both groups is carried out between 08:00 and 16:00 and the body weights of the infants are measured daily with the same scale before feeding.The amount in which the food (breast milk) is prepared to be given orally to the baby is recorded. The feeding time of all infants was limited to a maximum of 30 minutes. The feeding time of the infants are recorded in the feeding follow-up form. Before, during and after feeding, the heart rate, SPO2 and respiratory rates of the infants are recorded by pulse oximetry. During feeding, infants are evaluated with their early feeding skills by an observing nurse and their scores are recorded. Physiological parameters of infants are recorded before, during and after feeding is started, infants who are desaturated (SPO2 below 90%) during feeding are rested and feeding is continued after their saturation rises above 90% and these rest periods are also included in the feeding. After the decision to switch to oral feeding, the infants in the experimental group are fed 3 meals a day with the supplemental feeding system (daytime feedings), other meals are carried out with a bottle, and all the feedings of the infants in the control group are carried out with a bottle, which is the service routine. Infants' nutritional skills are evaluated at each meal, and their physiological measurements are recorded. After the evaluations of the infants who could not take the whole recommended amount of food in both groups (feeding time, recommended amount of food, amount of food the infant took, early feeding skill score and physiological parameters were recorded, the nurse completes the feeding of the infant with a bottle. The infants are followed up between 8-16 hours. The evaluations made at 3 meals are recorded. Infants who are fed orally for 8 meals a day for two consecutive days, and who can take 80% of the amount of food given at each meal, are considered to have switched to full oral feeding and the follow-up of the ınfants are stopped. The study followed the CONSORT guideline for reporting randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Postmenstrual age between 34-36 weeks (preterm babies at 34 and 36 weeks of gestation will be included),
* Over 1500 g,
* Switching to oral feeding after feeding with orogastric tube,
* Breastfed during gavage feeding,
* Those who have not completed the first 24 hours in the transition from orgastric tube feeding to the oral feeding process,
* Having cues of readiness for feeding (tolerating enteral nutrition, having a stable oxygen saturation and respiration during feeding, having the ability to lick, swallow and suck, react when mouth and lip are given stimuli),
* The mother's willingness to breastfeed her baby,
* Preterm infants of parents who volunteered to participate in the study will be included.

Exclusion Criteria:

* Having diseases other than being preterm,
* Capable of successfully taking the breast at the first attempt (Early Feeding Skill/EFS: 57),
* With congenital anomaly,
* With chromosomal disorders,
* With sepsis,
* With intracranial bleeding,
* Those with a very low birth weight below 1500 g and
* Preterm babies younger than 34 weeks of gestation will be excluded.

Ages: 34 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Early Feeding Skills | through study completion, an average of 10 days
  Before, during and after three feedings between 08:00 and 16:00

SECONDARY OUTCOMES:
Physiological parameters 1 (peak heart rate/minute) | through study completion, an average of 10 days
  Before, during and after three feedings between 08:00 and 16:00
Physiological parameters 2 (oxygen saturation/ %) | through study completion, an average of 10 days
  Before, during and after three feedings between 08:00 and 16:00
Physiological parameters 3 (respiratory rate/minute) | through study completion, an average of 10 days
  Before, during and after three feedings between 08:00 and 16:00

CONTACTS AND LOCATIONS:
Overall Officials: Fatma BOZDAĞ, Lecturer, Principal Investigator — Harran University
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No